CLINICAL TRIAL: NCT04517279
Title: Advancing the Early Psychosis Intervention Network in Texas
Brief Title: Peer Approaches to Substances in Early Psychosis Programs: A Pilot Study of a Peer-Led Intervention
Acronym: PAS-EPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Southern Methodist University (Other); Indiana University (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Molly Lopez, Research Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MH120599 (NIH)
Record Dates: First submitted 2020-08-12; First posted 2020-08-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Psychotic Disorders; Substance Use
Keywords: early psychosis; cannabis use; alcohol use; substance use
MeSH Terms: conditions — Psychotic Disorders; Substance-Related Disorders; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: The model is a cluster randomized controlled trial with randomization at the team level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Approaches to Substances in Early Psychosis Programs (Experimental): The Peer Approaches to Substances in Early Psychosis Programs arm is an intervention focused on enhancing the recovery capital of individuals in early psychosis care. The intervention is provided by a peer provider, operating on the coordinated specialty care team
  Interventions: Behavioral: Peer Approach to Substances in Early Psychosis Programs
- Usual Care (Active Comparator): The peer providers operating under the Usual Care condition will continue to provide peer support services to individuals within the coordinated specialty care team.
  Interventions: Behavioral: Usual Care Peer Services

INTERVENTIONS:
Behavioral: Peer Approach to Substances in Early Psychosis Programs — The intervention is consists of four core practice domains. Domain one includes practices that explore a young person's perspective, experience and beliefs around substances, validate through sharing personal experiences, and connect the young person with information around substances to inform decision-making. Domain two includes activities that support goals around substance use, including exploring motivation to change, identifying available supports, and planning to reduce negative effects of substance use. Domain three includes strategies to build recovery capital, such as enhanced social support. Domain four includes advocacy strategies within the CSC team to support client engagement and team coordination.
  Arms: Peer Approaches to Substances in Early Psychosis Programs
Behavioral: Usual Care Peer Services — Usual peer services involves supporting the process of change for individuals with mental health disorder to improve their health and wellness, live a self-directed life, and strive to reach their full potential.
  Arms: Usual Care

SUMMARY:
The aim of the study is to pilot a peer-provided, manualized intervention to increase the proportion of young people with first episode psychosis who reduce or stop substance use and improve psychiatric and functional outcomes. Coordinated specialty care teams will be randomly assigned to implement the intervention, Peer Approaches to Substances in Early Psychosis Programs (PAS-EPP), or usual care. The pilot study aims to: (a) determine if peer providers can implement PAS-EPP with adequate fidelity; (b) determine if youth and young adults engage in the intervention with peer providers and find it acceptable; (c) estimate the rates of drop-out for each of the two study arms; (d) estimate both between-participant (within-provider team) and between-team variability on key outcome measures; and (e) identify any changes needed to the intervention approach, manual, or training materials. The pilot study will set the stage for a future comparative cluster randomized trial of the intervention;

DETAILED DESCRIPTION:
The pilot study examines the feasibility of a cluster randomized controlled trial to measure the effectiveness of Peer Approaches to Substances in Early Psychosis Programs (PAS-EPP) compared to usual care (UC). PAS-EPP is a peer-led, manualized intervention to support youth and young adults receiving treatment for early psychosis with reducing or stopping problematic substance use. Peer providers, who represent clusters of service participants, will participate in a one-day PAS-EPP training. Training will include exploring the theoretical basis for the intervention approach and logic model, impact of service participant and peer provider on intervention design, the intervention strategies, and opportunities to build skill in each intervention component (e.g., role play with feedback). Peer providers will also receive monthly supervision to support intervention fidelity and resolve questions.

The proposed pilot study aims to: (a) determine if peer providers can implement PAS-EPP with adequate fidelity; (b) determine if youth and young adults engage in the intervention with peer providers and find it acceptable; (c) estimate the rates of drop-out for each of the two study arms; (d) estimate both between-participant (within-provider team) and between-team variability (e.g., standard deviation, interquartile range) on key outcome measures for a future comparative cluster randomized trial of the intervention; and (e) identify any changes needed to the intervention approach, manual, or training materials.

Twenty-five teams across 15 sites will be randomly assigned to PAS-EPP or UC, ensuring that the three sites with more than one team have at least one team randomized to each arm. All youth meeting eligibility criteria will be enrolled in the study and will receive either PAS-EPP or UC, based on the assignment status of their provider team. Intervention integrity will be measured through a peer-completed fidelity checklist. Participant outcomes will be measured through existing data collection at each participating organization. All participant outcome and service data is reported through the EPINET-TX platform, which allows for measurement-based care at participating sites and research using de-identified data.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in a CSC program during the defined study period;
* continued program enrollment at six month follow-up from program entry;
* continued alcohol/substance use at six-month follow-up from program entry.

Exclusion Criteria:

* none

Ages: 15 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Alcohol Use | 6 months after initiation of the intervention
  The primary outcome is the use of alcohol within the past 6 months as measured by the Alcohol Use Scale. The scale ranges from 1 to 5, with higher scores indicating more significant severity. Alcohol use is measured by a score of 2 or greater.
Alcohol Use | 12 months after initiation of the intervention
  The primary outcome is the use of alcohol within the past 6 months as measured by the Alcohol Use Scale. The scale ranges from 1 to 5, with higher scores indicating more significant severity. Alcohol use is measured by a score of 2 or greater.
Drug Use | 6 months after initiation of the intervention
  The primary outcome is the use of substances within the past 6 months as measured by the Drug Use Scale. The scale ranges from 1 to 5, with higher scores indicating more significant severity. Drug use is measured by a score of 2 or greater.
Drug Use | 12 months after initiation of the intervention
  The primary outcome is the use of substances within the past 6 months as measured by the Drug Use Scale. The scale ranges from 1 to 5, with higher scores indicating more significant severity. Drug use is measured by a score of 2 or greater.
Role Functioning | 6 months after initiation of the intervention
  The primary outcome is measured on the Global Functioning: Role scale (current). The scale ranges from 0 to 10, with higher scores reflecting better role functioning.
Role Functioning | 12 months after initiation of the intervention
  The primary outcome is measured on the Global Functioning: Role scale (current). The scale ranges from 0 to 10, with higher scores reflecting better role functioning.
Social Functioning | 6 months after initiation of the intervention
  The primary outcome is measured on the Global Functioning: Social scale (current). The scale ranges from 0 to 10, with higher scores reflecting better role functioning.
Social Functioning | 12 months after initiation of the intervention
  The primary outcome is measured on the Global Functioning: Social scale (current). The scale ranges from 0 to 10, with higher scores reflecting better role functioning.

SECONDARY OUTCOMES:
Stage of Change | 6 months after initiation of the intervention
  This secondary outcome is measured on the Substance Abuse Treatment Scale. The scale is ordinal, with 1 reflecting the "pre-engagement" stage and 7 reflecting "relapse prevention." Higher numbers reflect a more advanced stage of substance use treatment.
Stage of Change | 12 months after initiation of the intervention
  This secondary outcome is measured on the Substance Abuse Treatment Scale. The scale is ordinal, with 1 reflecting the "pre-engagement" stage and 7 reflecting "relapse prevention." Higher numbers reflect a more advanced stage of substance use treatment.
Perceived Well-being | 6 months after initiation of the intervention
  This secondary outcome is measured by the Personal Well-being Inventory. The summary score ranges from 0 to 100, with higher scores reflecting greater subjective well-being.
Perceived Well-being | 12 months after initiation of the intervention
  This secondary outcome is measured by the Personal Well-being Inventory. The summary score ranges from 0 to 100, with higher scores reflecting greater subjective well-being.
Recovery | 6 months after initiation of the intervention
  This secondary outcome is measured by the Questionnaire about the Process of Recovery. The total score ranges from 0 to 60, with higher scores reflecting greater recovery.
Recovery | 12 months after initiation of the intervention
  This secondary outcome is measured by the Questionnaire about the Process of Recovery. The total score ranges from 0 to 60, with higher scores reflecting greater recovery.
Severity of Psychiatric Symptomatology | 6 months after initiation of the intervention.
  This secondary outcome is measured by the Brief Psychiatric Rating Scale. The total score ranges from 0 to 108, with higher scores reflecting greater severity.
Severity of Psychiatric Symptomatology | 12 months after initiation of the intervention.
  This secondary outcome is measured by the Brief Psychiatric Rating Scale. The total score ranges from 0 to 108, with higher scores reflecting greater severity.

OTHER OUTCOMES:
Participant qualitative feedback | 12 months after initiation of the intervention.
  Some participants will participate in qualitative interviews on acceptability of the intervention.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Integral Care, Austin, Texas
  - Spindletop Centers, Beaumont, Texas
  - West Texas Centers, Big Spring, Texas
  - Metrocare Services, Dallas, Texas
  - Denton County MHMR, Denton, Texas
  - The Harris Center for Mental Health and IDD, Houston, Texas
  - Border Region Behavioral Health Center, Laredo, Texas
  - Community Healthcore, Longview, Texas
  - Burke, Lufkin, Texas
  - Coastal Plains, Portland, Texas
  - Bluebonnet Trails Community Center, Round Rock, Texas
  - Center for Healthcare Services, San Antonio, Texas
  - Central Counties Services, Temple, Texas
  - Andrews Behavioral Health, Tyler, Texas
  - Pecan Valley Centers, Weatherford, Texas

IPD SHARING:
Plan to Share IPD: Yes
Yes, data from this study will be submitted to the NIMH National Data Archive, along with appropriate data documentation.
Time Frame: The data is estimated to be available by 8/31/2026.
Access Criteria: The study data will be available to qualified researchers affiliated with an NIH-recognized institution through a request to the NIMH National Data Archive.
URL: https://nda.nih.gov/